CLINICAL TRIAL: NCT03989752
Title: Effects of an Overground Walking Program With Robotic Exoskeleton in Long-term Manual Wheelchair Users With a Chronic Spinal Cord Injury
Brief Title: Overground Walking Program With Robotic Exoskeleton in Long-term Manual Wheelchair Users With Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Collaborators: Université de Montréal (Other); Université du Québec a Montréal (Other)
Responsible Party: Principal Investigator, Dany H. Gagnon, Senior researcher, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DG-SO-18A
Record Dates: First submitted 2019-06-07; First posted 2019-06-18 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Spinal Cord Injuries
Keywords: Assistive Technology; Locomotion; Rehabilitation; Robotics
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable robotic exoskeleton-assisted walking program (Experimental): Total of 34 training sessions (60 min/session) during 16 weeks (1-3 session/week). Session intensity will be individualized and safely progressed thereafter (standing time, number of steps) to maintain a moderate-to-vigorous intensity (Borg rate of perceived exertion ≥12/20).
  Interventions: Device: Wearable Robotic Exoskeleton for Ambulation

INTERVENTIONS:
Device: Wearable Robotic Exoskeleton for Ambulation — 16-week walking program (34 sessions) with an overground walking robotic exoskeleton guided by a certified physical therapist

SUMMARY:
Many individuals with a spinal cord injury (SCI) use a wheelchair as their primary mode of locomotion. The prolonged non-active sitting time associated to this mode of locomotion contributes to development or worsening of numerous adverse health effects affecting musculoskeletal, endocrino-metabolic and cardiorespiratory health. To counter this vicious circle, engaging in a walking program with a wearable robotic exoskeleton (WRE) is a promising physical activity intervention. This study aims to measure the effects of a WRE-assisted walking program on musculoskeletal, endocrino-metabolic and cardiorespiratory health.

DETAILED DESCRIPTION:
Many individuals with a spinal cord injury (SCI) rely on manually propelled wheelchairs as their primary source of locomotion, leading to increased non-active sitting time, reduced physical activity and reduced lower extremity (L/E) weight bearing. This contributes to the development or worsening of complex and chronic secondary health problems, such as those affecting musculoskeletal (e.g., osteoporosis), endocrine-metabolic (e.g., hypertension, dyslipidemia, type 2 diabetes) and cardiorespiratory (e.g., poor aerobic fitness) health. Ultimately, these health problems may negatively affect functional capabilities and reduce quality of life.

Preliminary evidence has shown that engaging in a walking program with a wearable robotic exoskeleton (WRE) is a promising intervention. In fact, WRE-assisted walking programs promote L/E mobility and weight bearing (a crucial stimulus for maintaining bone strength in individuals with SCI), while also soliciting the trunk and upper extremity muscles and cardiorespiratory system.

This study aims to measure the effects of a WRE-assisted walking program on 1) bone strength, bone architecture and body composition, 2) endocrino-metabolic health profile and 3) aerobic capacity.

Twenty (20) individuals with a chronic (> 18 months) SCI will complete 34 WRE-assisted training sessions (1 h/session) over a 16-week period (1-3 sessions/week). Training intensity will be progressed (i.e., total standing time, total number of steps taken) periodically to maintain a moderate-to-vigorous intensity (≥ 12/20 on the Borg Scale). All training sessions will be supervised by a certified physical therapist.

Main outcomes will be measured one month prior to initiating the WRE-assisted walking program (T0), just before initiating the WRE-assisted walking program (T1), at the end of the WRE-assisted walking program (T2) and two months after the end of the WRE-assisted walking program (T3).

Descriptive statistics will be used to report continuous and categorical variables. The alternative hypothesis, stipulating that a pre-versus-post difference exists, will be verified using Repeated Mesures ANOVAs or Freidman Tests.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic or non-traumatic spinal cord injury between C6 and T10 neurological level at least 18 months pre-enrollment
* Long-term wheelchair use as primary means of mobility (non-ambulatory)
* Normal cognition (Montreal Cognitive Assessment Score ≥26/30)
* Understand and communicate in English of French
* Reside in the community within 75 km of the research site

Exoskeleton-specific inclusion criteria:

* Body mass ≤100 kg
* Height=1.52-1.93 m
* Pelvis width=30-46 cm
* Thigh length=51-61.4 cm
* Lower leg length=48-63.4 cm
* Standing tolerance ≥30 minutes with full lower extremity weight-bearing

Exclusion Criteria:

* Other neurological impairments aside from those linked to the spinal cord injury (e.g., severe traumatic brain injury)
* Concomitant or secondary musculoskeletal impairments (e.g., hip heterotopic ossification)
* History of lower extremity fracture within the past year
* Unstable cardiovascular or autonomic system
* Pregnancy
* Any other other conditions that may preclude lower extremity weight-bearing, walking, or exercise tolerance in the wearable robotic exoskeleton

Exoskeleton-specific exclusion criteria:

* Inability to sit with hips and knees ≥90° flexion
* Lower extremity passive range of motion limitations (hip flexion contracture ≥5°, knee flexion contracture ≥10°, and dorsiflexion ≤-5° with knee extended)
* Moderate-to-sever lower extremity spasticity (>3 modified Ashworth score)
* Length discrepancy (≥1.3 or 1.9 cm at the thigh or lower leg segment)
* Skin integrity issues preventing wearing the robotic exoskeleton

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Change in bone mass density (BMD) and architecture in the lower extremity | One month prior to intiating the walking program (T0), baseline at the initiation of the walking program (T1), at the end of the walking program (T2), two months after the end of the walking program (T3)
  Areal BMD will be calculated with dual-energy X-ray absorptiometry (DXA) at the proximal tibial plateau, distal femur, femoral neck and the 1st to the 4th lumbar vertebrae. Volumetric BMD and microarchitecture parameters of the trabecular and cortical bones (mineral content, mineral density, cross-sectional area, cortical thickness) at the distal femur and proximal tibia will be captured with peripheral quantitative computed tomography (pQCT).
Change in body composition | One month prior to intiating the walking program (T0), baseline at the initiation of the walking program (T1), at the end of the walking program (T2), two months after the end of the walking program (T3)
  DXA scans will be used to quantify total and regional body fat and fat free tissue mass (and relative percentages).
Change in muscle size | One month prior to intiating the walking program (T0), baseline at the initiation of the walking program (T1), at the end of the walking program (T2), two months after the end of the walking program (T3)
  Cross-sectional images of the radius, tibia and femur captured with pQCT will be used to measure muscle cross-sectional area.
Change in intramuscular fat infiltration | One month prior to intiating the walking program (T0), baseline at the initiation of the walking program (T1), at the end of the walking program (T2), two months after the end of the walking program (T3)
  Cross-sectional images of the radius, tibia and femur captured with pQCT will be used to measure intramuscular fat infiltration (i.e., muscle density).

SECONDARY OUTCOMES:
Change in bone turnover biomarkers | One month prior to intiating the walking program (T0), baseline at the initiation of the walking program (T1), at the end of the walking program (T2)
  Bone turnover (i.e., serum procollagen type I N-terminal peptide (P1NP), serum C-terminal cross-linking telopeptide (β-CTX) and 25-hydroxyvitamin D) biomarkers will be quantified using fasting blood samples.
Change in glycemic biomarkers | One month prior to intiating the walking program (T0), baseline at the initiation of the walking program (T1), at the end of the walking program (T2)
  Glycemic (i.e., fasting glucose, insulin, glycosylated hemoglobin (Hb A1C)) biomarkers will be quantified using fasting blood samples.
Change in insulin resistance | One month prior to intiating the walking program (T0), baseline at the initiation of the walking program (T1), at the end of the walking program (T2)
  Insulin resistance (hemeostatic model assessment (HOMA-1R)) will be quantified using fasting blood samples.
Change in lipide profile | One month prior to intiating the walking program (T0), baseline at the initiation of the walking program (T1), at the end of the walking program (T2)
  Lipid (i.e. Total cholesterol, HDL, LDHL, tryglicerides, ApoB) biomarkers will be quantified using fasting blood samples.
Change in inflammatory biomarkers | One month prior to intiating the walking program (T0), baseline at the initiation of the walking program (T1), at the end of the walking program (T2)
  Inflammatory (hsC-reactive protein, TNF-alpha, interleuken-6) biomarkers will be quantified using fasting blood samples.
Change in aerobic capacity | Baseline at the initiation of the walking program (T1), at the end of the walking program (T2)
  The Six-minute wheelchair propulsion test will be preformed with continuous expiratory gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dany H. Gagnon, PT, PhD, Principal Investigator — Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Locations (1):
- Institut universitaire sur la réadaptation en déficience physique de Montréal (IURDPM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data that underlie the results submitted for publication in peer-reviewed journal (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement
URL: http://crir.ca

REFERENCES:
- [Derived] Bass A, Morin SN, Guidea M, Lam JTAT, Karelis AD, Aubertin-Leheudre M, Gagnon DH; Montreal Exoskeleton Walking Program (MEWP) Group. Potential Effects of an Exoskeleton-Assisted Overground Walking Program for Individuals With Spinal Cord Injury Who Uses a Wheelchair on Imaging and Serum Markers of Bone Strength: Pre-Post Study. JMIR Rehabil Assist Technol. 2024 Jan 1;11:e53084. doi: 10.2196/53084. PMID 38163294
- [Derived] Bass A, Aubertin-Leheudre M, Vincent C, Karelis AD, Morin SN, McKerral M, Duclos C, Gagnon DH. Effects of an Overground Walking Program With a Robotic Exoskeleton on Long-Term Manual Wheelchair Users With a Chronic Spinal Cord Injury: Protocol for a Self-Controlled Interventional Study. JMIR Res Protoc. 2020 Sep 24;9(9):e19251. doi: 10.2196/19251. PMID 32663160